CLINICAL TRIAL: NCT02795728
Title: Fuji Type VII Sealants Versus Resin Based Sealants. A Clinical Trial
Brief Title: Fuji Type VII Sealant Versus Resin Based Sealant. A Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kamineni Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr. Praveen B.H, Assistant Professor, Kamineni Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSCDS
Record Dates: First submitted 2016-05-28; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Fuji type VII is a GIC based sealant with an additional property of high fluoride release
  Interventions: Other: Application of the GIC based sealant
- Resin based sealant (Active Comparator): Helioseal F is a resin based sealant
  Interventions: Other: Resin based sealant

INTERVENTIONS:
Other: Application of the GIC based sealant — Application of the GIC based sealant was carried out according to the manufacturer's instructions.
  Arms: Experimental arm
Other: Resin based sealant — Application of the resin based sealant on the occlusal surfaces was carried out as per the manufacturer s recommendations.
  Arms: Resin based sealant

SUMMARY:
Purpose: To evaluate the retention and caries preventive effect of the glass-ionomer fissure sealants and resin-based fissure sealant. Materials and Methods: Using a split mouth design ,a double blind randomized controlled clinical trial was conducted to compare the retention and the caries preventive effect of light cure resin base sealant (3M ESPE) and Glass ionomer sealant (FUJI). The study comprised of 120 government school children of 7-9 years age group. The glass-ionomer sealant and resin-based sealant were applied randomly on either side of the first mandibular permanent molars. They were recalled for assessment of sealant retention at intervals of 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children with a fully erupted contra lateral permanent mandibular first molars with well-defined deep pits and fissures and molars free of mucosal tissue are included in the study.

Exclusion Criteria:

* Molars with developmental anomalies, hypoplastic teeth were promptly excluded

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Retention of the sealant | Baseline to 1 year
  Retention of the sealants will be assessed by using the Simensons criteria

SECONDARY OUTCOMES:
Caries incidence | Baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prathibha Rao, MDS, Study Director — Sri Sai college of Dental surgery
Locations (1):
- Sri Sai college of Dental surgery, Vikārābād, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes